CLINICAL TRIAL: NCT02200367
Title: AN e- MENTAL HEALTH COLLABORATIVE PROGRAMME TO DEPRESSION MANAGEMENT IN RURAL PRIMARY CARE IN CHILE:A PILOT CLINICAL STUDY.
Brief Title: E-mental Health Support for Rural Areas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government)
Responsible Party: Principal Investigator, Graciela Rojas Castillo, Dr.med. Psychyatrist, University of Chile
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1100205
Record Dates: First submitted 2014-07-15; First posted 2014-07-25 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Depression
Keywords: Primary health care; Computer communication network; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- e-mental health collaborative programme (Experimental): It is a complex intervention to support primary care providers of rural primary care service to manage depressed patients. Primary care providers at the intervention sites were supported by psychiatrist using an electronic platform.Patients were monitored through a call center.
  Interventions: Behavioral: e-mental health collaborative programme
- Usual Care (Other): Patients in this arm received all the interventions that are guaranteed for the persons with depression in Chile: treatment in the primary clinics with the primary care team and referral to the regional specialized psychiatric service
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: e-mental health collaborative programme
  Arms: e-mental health collaborative programme
Other: Usual Care
  Arms: Usual Care

SUMMARY:
In the treatment of depression, primary care team play an important role, but they are most effective when inserted into a collaborative model of disease management.

Hypotheses:Depressed patients treated in rural primary care clinics participating in a e-mental heath collaborative programme to manage depression achieve at least 20% better recovery rates in comparison with the control group three months after the baseline assessment.

Goal: to compare the effectiveness of a e-mental health collaborative programme with usual care in rural primary-care clinics.

Methodology: a clinical trial with two arms will be conducted in 13 community rural hospitals in Chile. The active group will participate in a collaborative programme between primary care teams and specialized teams, with support from an electronic platform and a call center.The control group will receive usual care, according to the Ministry of Health's Guidelines to Depression.To evaluate inclusion criteria -depressive patients aged between 18 and 70 years- and exclusion criteria -current in treatment for depression- an interview will be used that will include the Mini-International Neuropsychiatric Interview (MINI) to evaluate depression .The principal outcome will be depressive symptoms measured with the Beck Depression Inventory (BDI-I), and secondary outcome quality of life measured with the Health Survey (SF-36) at three and six months after baseline assessment.To detect a difference of 20%, in a one-sided model, with an alpha of 5% and power of 80%, would require 152 depressed persons (76 to intervention and 76 to control group).A design effect of 1.35 based on an Intraclass Coefficient Correlation (ICC) of 0,03839 and 13 clinics were considered. After applying the design effect the sample needed increased to 206 depressed persons. Considering a retention rate of approximately 85% 237 depressed cases will be needed.

A program of this kind may be useful to assist primary care teams in remote areas of the country, in order to improve treatment outcomes for depression that is currently addressed at the primary care level.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 or more with a current major depressive episode according to Diagnostic and Statistical Manual of Mental Disorders IV criteria (DSM-IV)

Exclusion Criteria:

* Depressive treatment currently in process.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2011-01; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Depressive Symptoms change after baseline | three and six months
  BDI-I

SECONDARY OUTCOMES:
Quality of Life change after baseline | three and six months
  SF-36

REFERENCES:
- [Derived] Rojas G, Guajardo V, Martinez P, Castro A, Fritsch R, Moessner M, Bauer S. A Remote Collaborative Care Program for Patients with Depression Living in Rural Areas: Open-Label Trial. J Med Internet Res. 2018 Apr 30;20(4):e158. doi: 10.2196/jmir.8803. PMID 29712627